CLINICAL TRIAL: NCT05244863
Title: The Relationship of Proximal and Distal Muscle Strength With Upper Extremity Functional Skills in Geriatric Individuals With Essential Tremor
Brief Title: The Relationship of Muscle Strength With Functional Skills in Geriatric Individuals With Essential Tremor
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Zekiye İpek KATIRCI KIRMACI, Asst. Prof., Kahramanmaras Sutcu Imam University
Other Study IDs: zipekkatirci
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Essential Tremor
Keywords: muscle strength; Geriatric individuals; Functional manual dexterity
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- One group: Geriatric individuals
  Interventions: Other: Test

INTERVENTIONS:
Other: Test — Measurements

SUMMARY:
Essential tremor is one of the most common movement disorders in the world and is characterized by postural and/or kinetic tremor.

Although the prevalence studies show differences due to the absence of a biological marker of the disease, it has been shown that the disease affects 4% of the population over 40 years of age and this rate may increase up to 14% in the population over 65 years of age. The annual incidence of Essential Tremor was found to be 616 per 100 thousand.

The incidence of the disease increases with age. An incidence study shows that the disease increases progressively with age, with a sharp increase after age 49. In another study, it was stated that the age of onset of the disease showed a bimodal distribution, reaching the highest level in the second and sixth decades. It is stated that the severity and disability of tremor increase with age. The female-to-male ratio of the disease was found to be equal, but it was shown that more head tremor developed in females.

Although the factors affecting essential tremor are aging, stress, family history, excessive caffeine consumption, smoking, muscle weakness, distal and proximal muscle strength differences were detected in young individuals with tremor. The aim of this study was to investigate the relationship between proximal and distal muscle strength and upper extremity functional skills in geriatric individuals with essential tremor.

DETAILED DESCRIPTION:
In order for many elderly individuals to maintain their independence in functional activities, it is critical that the upper extremity dexterity is at a good level. Because the upper extremity needs to be functional in the realization of social relations such as writing, cooking, combing their hair, brushing their teeth, and participating in recreational activities. Due to the importance of maintaining functional independence in old age, many reviews have attempted to identify primary age-related neuromuscular changes that have an impact on the decreased function of most of the elderly. Age-related declines in function can be explained by increased motor unit firing rate variability of various central and peripheral nervous systems. It is thought to increase tremor in the altered synchronization between motor units in agonist and antagonist muscles, as well as impaired activation between agonist and antagonist muscles. Muscle strength differences in upper extremity functional skills were detected between proximal and distal muscle groups in young individuals with Essential Tremor. In a study investigating the effect of resistance exercise training on tremor in geriatrics, the changes in postural tremor with resistance training in healthy older adults were investigated. In this study; The frequency and severity of tremor of two different groups that received strength and coordination training were evaluated, and it was stated that there was a significant difference in the strength training group.

In this study, which is the only literature study in which strength training was applied to geriatric individuals with essential tremor, it was not specified on which muscle groups the strength training would be effective. In our study, determining the strength differences of the proximal and distal muscle groups of geriatric individuals with essential tremor will enable the creation of effective programs specific to the individual and muscle groups in the rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary geriatric individuals aged 60-85 years with and without tremor
* with a mini mental test score above 24,

Exclusion Criteria:

* have diabetic neuropathy
* have undergone hand surgery
* upper and lower motor paralysis
* a history of hand fracture

Ages: 60 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: geriatric individuals with and without tremor
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
ahn-Tolosa-Marin Tremor Rating Scale | At baseline
  It is a widely used clinical assessment scale for tremor. The severity of tremor body parts is determined as 5 grades from 0 (absent) to 4 (severe)
Proximal muscle strength | At baseline
  Digital dynamometer was used to evaluate muscle strength.
Dİstal muscle strength | At baseline
  Jamar dynamometer was used to evaluate muscle strength.
Disability Arm Shoulder Hand | At baseline
  The DASH-T questionnaire is completed by the individual and consists of 3 parts: the functional/symptom (DASH-FS), the business model (DASH-W), and the sports-musicians model (DASH-SM). The person answers all questions according to a 5-point Likert system (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: not able to do at all). A score between 0-100 is obtained from each section. The higher the score, the higher the disability.
Nine Holes Peg test | At baseline
  The test is performed with the patient in a sitting position. The patient is asked to line up the nine sticks inside the box on the table as quickly as possible into the holes of the other box, and remove them immediately after finishing. The test is started with the dominant hand, the time is measured with a stopwatch, and it is started when the hand touches the bars and ends when the last stick is placed in the box.

CONTACTS AND LOCATIONS:
Overall Officials: Zekiye İpek Katırcı Kırmacı, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaraş Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided